CLINICAL TRIAL: NCT02258880
Title: A Phase 2, Multicenter, Multinational, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of SUN13837 Administered 28 Doses (27/28 Days) to Adult Subjects With an Acute Ischemic Stroke
Brief Title: Efficacy, Safety, Tolerability and Pharmacokinetics of SUN13837 to Treat Acute Stroke
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: study was stopped for business/administrative reasons and not for patient safety concerns
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASBI 802
Record Dates: First submitted 2014-09-29; First posted 2014-10-08 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Stroke
Keywords: Acute Stroke; Outcome Measures; Physical Performance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SUN13837 (Experimental): Drug: SUN13837 daily for 28 days.
  Interventions: Drug: SUN13837
- Placebo (Placebo Comparator): Placebo: Matching Placebo daily for 28 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SUN13837
  Arms: SUN13837
Drug: placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of SUN13837 and to determine whether SUN13837 improves the physical performance, relative to placebo, following an acute stroke in adult subjects.

ELIGIBILITY:
Each subject must meet all of the following criteria to participate in the study:

1. Male or female subjects between 18 and 85 years, inclusive
2. Subjects with no prior history of stroke (unless the stroke was not associated with a motor deficit)
3. Subjects must score at least 16 points on the standard MMSE during baseline assessments
4. Subjects must have a total score between 7 and 30, inclusive, out of 35 on the S-STREAM administered between 24 and 48 hours after the onset of acute stroke
5. Subjects must have an estimated pre-stroke mRS of 0 or 1
6. Male subjects agree to be heterosexually abstinent or use appropriate contraception
7. Female subjects must have undergone menopause or, if premenopausal, must have a negative pregnancy test at baseline. Female subjects of childbearing potential agree to be sexually abstinent or must be willing to utilize adequate contraception
8. Subjects must be willing to provide verbal/nonverbal informed consent indicating voluntary consent to participate in the study (if a subject is unable to provide informed consent, but able to comply with other study procedures, the subject's LAR may provide consent)

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. Prior exposure to SUN13837
2. History of severe allergic reaction, whether explained or not, requiring a visit to the ER and/or medical intervention with epinephrine
3. Development of hemodynamic instability following the acute stroke
4. History of dementia, advanced Parkinson's disease, other significant movement disorders, or other clinically significant diseases which would jeopardize the safety of the subject or impact the validity of the study results
5. Presence of significant global or receptive aphasia
6. Presence of clinically significant abnormal laboratory values at the time of presentation in the ER
7. History of malabsorption or any gastrointestinal abnormality that could impair oral absorption
8. Finding of Grade 3 or 4 proliferative retinopathy on routine fundoscopic examination or history of proliferative retinopathy (Grade 3 or 4) in subjects with diabetes mellitus
9. Unable, as determined by the investigator, or unwilling to discontinue use of potent cytochrome (CYP) P450 3A4/5 inhibitors, potent CYP2D6 inhibitors, CYP3A inducers, or potent P glycoprotein (P gp) inhibitors
10. Current participation in another clinical study involving administration of an investigational product or history of such participation within 30 days of acute stroke onset

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in the Physical Performance Assessment in Stroke (PPAS) | 84 days

SECONDARY OUTCOMES:
The proportion of responders as measured by the PPAS | 84 days
Mean change from baseline in PPAS Patient Reported Outcome Subscale | 84 days
Mean change from baseline in Short Form-36 Physical Functioning Scale (SF-36 PF) | 84 days
Mean change from baseline in Gait Speed | 84 days
Proportion of responders as measured by the Modified Rankin Scale (mRS) | 84 days
Safety/Tolerability - Number of Participants with Adverse Events | 84 days

CONTACTS AND LOCATIONS:
Overall Officials: Ger Rikken, MD, Study Director — Asubio Pharmaceuticals, Inc.
Locations (47):
- United States (32):
  - Mobile, Alabama
  - Encinita, California
  - Oceanside, California
  - Sarasota, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Lexington, Kentucky
  - Marrero, Louisiana
  - New Orleans, Louisiana
  - Worcester, Massachusetts
  - Detroit, Michigan
  - Novi, Michigan
  - Southfield, Michigan
  - Kalispell, Montana
  - Reno, Nevada
  - Edison, New Jersey
  - Summit, New Jersey
  - Brooklyn, New York
  - Chapel Hill, North Carolina
  - Columbus, Ohio
  - Portland, Oregon
  - Bryn Mawr, Pennsylvania
  - Hershey, Pennsylvania
  - Paoli, Pennsylvania
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Chattanooga, Tennessee
  - Houston, Texas
  - Mechanicsville, Virginia
  - Midlothian, Virginia
  - Richmond, Virginia
- Canada (3):
  - Edmonton, Alberta
  - Victoria, British Columbia
  - Saint-Jérôme, Quebec
- Israel (6):
  - Haifa
  - Holon
  - Kfar Saba
  - Naharyia
  - Ramat Gan
  - Tel Aviv
- South Africa (6):
  - Bloemfontein, Free State
  - Alberton, Gauteng
  - Krugersdorp, Gauteng
  - Bellville, Western Cape
  - Somerset West, Western Cape
  - Worcester, Western Cape